CLINICAL TRIAL: NCT01093040
Title: A Phase I, Single-Center, Single-blind, Randomized, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Immunogenicity of CAT-354 Following Subcutaneous Administration in Healthy Male and Female Japanese Subjects
Brief Title: A Study to Assess the Safety and Immunogenicity of the Drug CAT-354 in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: MedImmune Ltd (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MI-CP224
Record Dates: First submitted 2010-03-19; First posted 2010-03-25 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
MeSH Terms: interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): CAT-354 will be administered by SC injection
  Interventions: Drug: CAT-354
- Cohort 2 (Experimental): CAT-354 will be administered by SC injection
  Interventions: Drug: CAT-354
- Cohort 3 (Experimental): CAT-354 will be administered by SC injection
  Interventions: Drug: CAT 354

INTERVENTIONS:
Drug: CAT-354 — 150 mg CAT-354 or placebo given SC on Day 1
  Arms: Cohort 1
Drug: CAT-354 — 300 mg CAT-354 or placebo given SC on Day 1
  Arms: Cohort 2
Drug: CAT 354 — 600 mg CAT-354 or placebo given SC on Day 1
  Arms: Cohort 3

SUMMARY:
To assess the safety of the administration of the drug (CAT-354) in healthy Japanese subjects.

DETAILED DESCRIPTION:
The study design allows a gradual escalation of dose with safety monitoring to ensure the safety of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 20 through 55 years at the time of screening
* Signed and dated written informed consent is obtained prior to any study related procedure taking place
* No significant abnormality on clinical examination or medical history (excluding atopic skin signs, symptoms and history)
* A normal 12-lead electrocardiogram (ECG) (no clinically significant abnormalities)
* Clinical chemistry, hematology and urinalysis results within the laboratory reference ranges or deemed not clinically significant by the Investigator
* A negative screen for drugs of abuse and alcohol
* The following reproductive criteria apply:
* Females(of child bearing potential) must have a negative pregnancy test prior to the dose of investigational product and, unless surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy), has a sterile male partner, or at least 2 years postmenopausal, or practices abstinence; must use 2 effective methods of avoiding pregnancy (including oral, transdermal, or implanted hormonal contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap with spermicide, or use of a condom with spermicide by the sexual partner) for 21 days prior to randomization, and must agree to continue using such precautions until 3 months after dosing with the investigational product; cessation of birth control after this point should be discussed with a responsible physician. A negative pregnancy test is required both at screening and prior to dosing.
* Males, unless surgically sterile, must use two effective methods of birth control with a female partner and must agree to continue using such contraceptive precautions from 21 days prior to randomization until 3 months after dosing with the investigational product.
* Japanese subjects. To be considered as 'Japanese', both of the subject's parents, and both sets of grandparents, must be Japanese. The subject must have been born in Japan, have a valid Japanese passport, and must not have lived outside Japan for more than 5 years.
* Body mass index (BMI) between 18 and 27 kg/m 2 , inclusive
* Able to comply with the requirements of the protocol

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Previously received monoclonal antibody, or a similar related protein, that might sensitize subjects to CAT-354 or to any component of the investigational product formulation
* History of an active infection within 4 weeks prior to screening, or evidence of clinically significant active infection, including ongoing chronic infection
* Any acute illness in the 14 days before Day 1 (Visit 2)
* Use of any medication (prescription or OTC) excluding hormonal contraception within 14 days (or 5-half lives, whichever is longer) of Day 1 dosing
* Involvement in another study of investigational medicinal product; within 2 months of the start of this study (Day 1) for small molecules, within 3 months of the start of this study for antibodies, or 5 half lives of the previously administered investigational product, whichever is the longer
* Any blood donation or significant loss of blood within 56 days of study initiation or plasma donation within 7 days of study initiation
* Subjects with immunodeficiency disorders
* Subjects who have a positive test for, or have been treated for hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* Any active concomitant disease including psychological disorders
* Subject is a participating Investigator, sub-Investigator, study coordinator, or employee of a participating Investigator, or is a first-degree relative of the aforementioned.
* Any factor which, in the opinion of the Investigator, would be associated with poor adherence to the protocol
* Female subjects: lactation

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety | Study Day 71
  The safety and tolerability of a single dose SC injection of CAT-354 in healthy male and/or female Japanese subjects will be assessed through the incidence of adverse events (AEs), and the assessment of vital signs, physical examinations, laboratory parameters, and electrocardiograms.

SECONDARY OUTCOMES:
Immunogenicity | Study Day 71
  The PK variables and IM variables of CAT-354 in healthy Japanese subjects will be evaluated. The incidence rate of positive serum antibodies to CAT-354 will be reported by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Katsuro Yagawa, M.D., Study Director — Astra Zeneca K.K.
Locations (1):
- Research Site, Glendale, California, United States